CLINICAL TRIAL: NCT06295718
Title: Tele-assessment of Functional Performance and Quality of Life in Patients With Duchenne Muscular Dystrophy: Validity and Reliability Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Sahra Şirvan (Other)
Responsible Party: Sponsor-Investigator, Sahra Şirvan, PhD Student, Istanbul University
Organization: Istanbul University (Other)
Other Study IDs: 2023/51
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy, Tele-assessment, Timed Performance Test, Quality of Life, Fatigue
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Fatigue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ambulatory Children with Duchenne Muscular Dystrophy: Participants who meet the inclusion criteria will be evaluated synchronously online using the Zoom platform in terms of the functional performance and quality of life parameters specified below, after ensuring the presence of a suitable environment and a stable internet connection. During the online evaluation, patients will be asked to perform the specified functions in front of the camera. In addition, the survey questions necessary to evaluate the quality of life will be expressed verbally to the participants. Inter-rater reliability will be examined by comparing the scores after being performed separately by two different physiotherapists. The reliability and validity of the online assessment will be investigated by repeating the same assessments online and face-to-face.
  * Timed Performance Tests
  * Upper Extremity Functions
  * Lower Extremity Functions
  * Quality of Life

SUMMARY:
Thanks to tele-assessment methods, it may be possible to evaluate DMD patients without traveling to clinical centers. In recent years, the applicability of remote assessment methods in DMD patients, as in many populations, is being investigated. However, studies have generally focused on a single evaluation parameter such as physical function, a special evaluation method or a special evaluation tool. The aim of this study is to investigate whether remote assessment of functional performance and quality of life in DMD patients is valid and reliable. If a valid and reliable tele-evaluation method that includes functional performance and quality of life parameters is found to be valid and reliable, the travel burden on patients and caregivers can be eased, patients' stress and anxiety related to travel can be reduced, caregivers can save time and energy and provide patients with the best possible treatment.

DETAILED DESCRIPTION:
DMD is a progressive muscle disease that causes difficulties in mobility and impairment of vital functions as a result of X chromosome-linked dystrophin deficiency. Symptoms appear between the ages of 3 and 5, and in untreated cases, loss of ambulation occurs around the age of 8-12. Long sitting periods due to wheelchair use increase the risk of contracture, osteopenia, fracture and scoliosis, and accompanying cardiorespiratory complications cause mortality in the early 20s in most cases. Determining functional performance in DMD is a guide for determining appropriate treatment options and objectively evaluating the effectiveness of treatment. However, the evaluation methods applied are performed in clinical environments that require frequent travel and require both time and physical effort. The aim of this study is to investigate whether remote assessment of functional performance and quality of life in DMD patients is valid and reliable. For this purpose, 20 volunteers diagnosed with DMD at Istanbul University-Cerrahpaşa Child Neurology Polyclinic and who meet the inclusion criteria will be evaluated in two ways, online and face-to-face, in terms of functional performance and quality of life parameters. In addition, scoring will be performed by two different physiotherapists during the evaluation and the reliability of the tele-evaluation among the evaluators will be examined. Functional performance timed performance tests, Brooke Upper Extremity Functional Classification and Vignos Lower Extremity Functional Classification; Quality of life will be evaluated with PedsQL-3.0 Neuromuscular Module and PedsQL Multidimensional Fatigue Scale. Thanks to valid and reliable tele-assessment methods for DMD patients, travel burden can be alleviated for both patients and caregivers, and disease-related stress and anxiety can be reduced. In this way, caregivers can save time and energy while providing the best care to patients.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Duchenne muscular dystrophy
* Being between the ages of 5-18
* Having ambulation skills
* Having internet access and technical requirements
* Having the ability to follow movement instructions
* Volunteering to participate in the study

Exclusion Criteria:

* Having cognitive or behavioral problems that may interfere with evaluation
* Having communication problems that may prevent evaluation
* Having a level of contracture that may prevent evaluation
* Having a systemic disease that may prevent evaluation

Ages: 5 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Male
Study Population: This research is a descriptive type observational study, and the population of the study will be 20 volunteer cases who were diagnosed with Duchenne Muscular Dystrophy at Istanbul University-Cerrahpaşa Faculty of Medicine Child Neurology Polyclinic and who meet the exclusion criteria. The study will be carried out at Istanbul University-Cerrahpaşa Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-03-02 (Estimated); Study Completion 2024-05-10 (Estimated)

PRIMARY OUTCOMES:
Timed Performance Tests | 2 days
  Timed performance tests are one of the frequently preferred outcome measures in patients with DMD. The time patients spend performing certain functions is recorded. The following functions will be evaluated in this study: • Getting up from the ground • Standing up from a chair • Don't wear a t-shirt • T-shirt removal • Collect 6 coins with one hand • Timed Up and Go Test
Brooke Upper Extremity Functional Classification (BUEFS) | 2 days
  Brooke Upper Extremity Functional Classification (BUEFS) will be used to evaluate the upper extremity functions of the cases. BUEFS is a valid, reliable and practical scale used to classify the upper extremity functions of individuals with DMD. It was developed by Brooke et al. in 1981. Individuals are classified between 1 and 6 according to the upper extremity activities they can perform, and higher stages indicate decreased functionality of the upper extremity.
Vignos Lower Extremity Functional Classification (VAEFS) | 2 days
  Vignos Lower Extremity Functional Classification (VAEFS) will be used to evaluate the lower extremity functions of the cases. VAEFS is a scale consisting of 10 stages that evaluates the level of ambulation in neuromuscular diseases. It was developed by Vignos et al. in 1963. Individuals are classified between 1 and 10 according to their ambulation level, and higher stages indicate a decrease in ambulation level. While the patient in the first stage can walk and climb stairs without support, in the highest stage he is bedridden.
PedsQL-3.0 Neuromuscular Module by PedsQL Multidimensional Fatigue Scale | 2 days
  The patients' quality of life will be evaluated using the PedsQL-3.0 Neuromuscular Module- the PedsQL Multidimensional Fatigue Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul University - Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No